CLINICAL TRIAL: NCT05233696
Title: Phase II Study of Radiotherapy in Combination With Chemotherapy and Immunotherapy in Patients With PD-L1-Positive Metastatic Triple-Negative Breast Cancer
Brief Title: Radiotherapy in Combo With Chemo and Immunotherapy in Patients With PD-L1 Positive Metastatic TNBC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-3117.cc
Record Dates: First submitted 2022-01-04; First posted 2022-02-10 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Triple Negative Breast Cancer; Locally Advanced Breast Cancer; Unresectable Breast Carcinoma; Metastatic Breast Cancer; PD-L1 Gene Mutation
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Paclitaxel; Radiotherapy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RT followed by nab-paclitaxel/paclitaxel plus pembrolizumab (Experimental): Nab-paclitaxel/paclitaxel plus pembrolizumab will be started within 7 days of completion of RT.
  Interventions: Drug: Nab-paclitaxel; Drug: Paclitaxel; Radiation: Radiation Therapy; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nab-paclitaxel — All patients are encouraged to receive nab-paclitaxel 100 mg/m2 IV D1 and D8 every 21 days (in combination with pembrolizumab) for at least 4-6 cycles per institutional standards and treating physicians' recommendations.
  Other Names: Abraxane
Drug: Paclitaxel — Paclitaxel can be substituted for nab-paclitaxel at the discretion of the treating physician 80 mg/m2 IV D1 and D8 every 21 days.
  Other Names: Abraxane
Radiation: Radiation Therapy — The treating radiation oncologist will select 1-4 sites of metastatic disease to target with radiation. All sites of disease may be targeted with radiation. Sites of metastatic disease planned to be biopsied should not be radiated.
Drug: Pembrolizumab — Patients will receive pembrolizumab 200 mg D1 every 21 days.
  Other Names: Keytruda

SUMMARY:
Patients with locally advanced unresectable or metastatic programmed cell death ligand (PD-L1) positive triple negative breast cancer (TNBC) will be treated with radiation to one-four sites of metastasis amenable to radiation (sites of disease to be selected at the discretion of the treating radiation oncologist) followed by initiation of systemic therapy with pembrolizumab plus nab-paclitaxel/paclitaxel. Patients will be treated with pembrolizumab plus nab-paclitaxel/paclitaxel within 7 days of completion of radiation. Repeat imaging of all sites of disease will be performed every 9 weeks and response will be assessed according to RECIST 1.1.

DETAILED DESCRIPTION:
Patients with locally advanced unresectable or metastatic PD-L1 positive TNBC will be treated with radiation to one-four sites of metastasis amenable to radiation (sites of disease to be selected at the discretion of the treating radiation oncologist) followed by initiation of systemic therapy with pembrolizumab plus nab-paclitaxel/paclitaxel. Patients will be treated with pembrolizumab plus nab-paclitaxel/paclitaxel within 7 days of completion of radiation. Repeat imaging of all sites of disease will be performed every 9 weeks and response will be assessed according to RECIST 1.1.

This is a two-stage, single-arm phase II study. Utilizing time-to-event outcomes, the investigators assumed an uninteresting 1-year PFS rate of 39% and a positive 1-year PFS rate of 60%. The first stage will enroll 17 subjects, with an additional 12 subjects to be enrolled in stage 2 if the trial is not stopped due to futility, for a total of 29 subjects. Enrollment will not be paused after the first stage of enrollment. At the time of the interim analysis the investigators would expect approximately 12 patients to have completed 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form including non-English speaking and non-reading participants.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Male or female aged ≥ 18 years.
4. Metastatic or locally advanced unresectable histologically documented TNBC as defined by absence of estrogen receptor (ER) and progesterone receptor (PR) expression and no HER2 amplification or over-expression by local pathology report.

   1. HER2 negativity is defined as either: in situ hybridization non-amplified (ratio of HER2 to CEP17 < 2 or single probe average HER2 gene copy number < 4 signals/cell OR IHC 0 or 1+).
   2. ER and PR negativity is defined as < 1% positive by IHC.
5. Treatment with < 1 prior line of systemic therapy in the metastatic setting or adjuvant/neoadjuvant setting if metastatic recurrence within 12 months of treatment.
6. Confirmed PD-L1 positive as defined by Combined Positive Score (CPS) > 10% by a CLIA-certified lab
7. At least one site of disease amenable to radiation therapy.
8. Clinically appropriate for treatment with nab-paclitaxel/paclitaxel plus pembrolizumab in the opinion of the treating investigator.
9. If the maximum number of non-biopsy subjects has accrued to the study, willingness to undergo 2 tumor biopsies and disease amenable to safe biopsy in the opinion of the treating investigator. NOTE: Tumor biopsies may be required, depending on the number of subjects who have agreed to undergo correlative studies.
10. Life expectancy of > 3 months per treating investigator.
11. ECOG performance status ≤ 1.
12. Baseline labs must meet the following criteria within 21 days of radiation initiation:

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
    2. Platelets ≥ 100,000/mcL.
    3. Hemoglobin ≥ 9.0 g/dL.
    4. Total bilirubin ≤1.5 x institutional upper limit of normal (ULN) or ≤ 3 x ULN for subjects with Gilbert's disease.
    5. AST (SGOT)/ALT (SGPT) ≤ 3 X institutional ULN or ≤ 5 X institutional ULN in liver metastasis are present.
    6. Serum creatinine < 1.5 X institutional ULN.
    7. INR and PTT < 1.5 X institutional ULN. This applies only to patients undergoing serial tumor biopsies.
13. All prior reversible treatment-related toxicities must have resolved to CTCAE v5.0 criteria of grade 1 or less (except alopecia).
14. Women must not be pregnant or breastfeeding.
15. Women of childbearing potential must have a negative pregnancy test before enrollment. Women who are not of childbearing potential defined as post- menopausal (amenorrheic for > 12 months) or undergone prior hysterectomy or bilateral salpingo-oophorectomy do not require pregnancy testing.
16. Willingness of male and females who are of childbearing potential to use medically acceptable contraception for the duration of the study, including 30 days after last dose of nab-paclitaxel/paclitaxel and 6 months after last pembrolizumab, whichever is longer. Male patients must refrain from donating sperm during these periods.
17. Availability of archival tumor tissue (core biopsy or surgical tumor blocks) for analysis. Sites will be asked to submit archival tissue (subjects may start the study if tissue is available at an outside hospital, but not yet requested or received).

Exclusion Criteria:

1. Any of the following interventions within the specified time frame prior to radiation:

   1. Radiation therapy within 21 days.
   2. Cytotoxic chemotherapy within 21 days (capecitabine within 14 days).
   3. Monoclonal antibodies within 21 days.
   4. Administration of an investigational agent that is not expected to be cleared prior to initiation of radiation.
2. More than one prior line of chemotherapy in the locally advanced unresectable or metastatic setting.
3. Prior treatment with a taxane in the metastatic setting. Prior taxane in the curative setting is allowed if treatment was completed ≥ 6 months prior to metastatic recurrence.
4. Prior receipt of immune checkpoint inhibitor (PD-L1, PD-1 or CTLA-4 inhibitors) less than 12 mos from metastatic recurrence.
5. Patients with active collagen vascular disease (CVD), specifically systemic lupus erythematosus or scleroderma. Patients with a history of CVD without evidence of active disease are eligible for enrollment at the discretion of the study PI.
6. History of immunodeficiency, hypersensitivity to pembrolizumab or other medical contraindication to receipt of immunotherapy.
7. Has active, or history of, pneumonitis requiring treatment with corticosteroids.
8. Has a known history of active tuberculosis.
9. Has a known history of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome - related illness (testing not required at screening).
10. Has known active hepatitis B (hepatitis B surface antigen reactive) or hepatitis C (qualitative HCV RNA is detected) (testing not required at screening).
11. Has received a live vaccine within 30 days prior to enrollment.
12. Has an active infection requiring treatment with oral or IV medication. Patients on antimicrobial, antifungal or antiviral prophylaxis are not specifically excluded if all other criteria are met.
13. Autoimmune disease that has required systemic treatment in the past 2 years (ie. with the use of disease modifying agents, systemic corticosteroids, or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
14. Symptomatic or uncontrolled central nervous system (CNS) metastases. Patients with treated brain metastasis with stable CNS imaging > 28 days after radiation and no requirement for corticosteroids are eligible.
15. Receipt of corticosteroid therapy at greater than physiologic dosing in the investigator's opinion within 14 days of the start of radiation therapy.
16. For patients undergoing serial tumor biopsies, known bleeding diathesis or history of abnormal bleeding or require anti-coagulation therapy that cannot be interrupted for biopsy.
17. Patients with a separate active cancer diagnosis for which the patient has not been without evidence of disease for at least 2 years.
18. Medical, psychiatric, cognitive or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the study protocol, or to complete the study.
19. Any severe concurrent disease or condition (including uncontrolled diabetes mellitus, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, or cardiac arrythmia) which, in judgment of the Investigator, would make the patient inappropriate for study participation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
1 year progression free survival rate | 36 months
  To determine the efficacy of radiotherapy in combination with chemotherapy plus immunotherapy as defined by 1-year PFS rate in patients with PD-L1-positive metastatic TNBC.

SECONDARY OUTCOMES:
Rate of in-field tumor control | 36 months
  In-field tumor control will be defined as stable disease (SD), partial remission (PR), or complete remission (CR), of the target lesion, by RECIST 1.1 criteria.
Determine overall response rate (ORR) | 36 months
  Determined by RECIST 1.1
Determine clinical benefit rate (CBR) | 36 months
  Defined as SD, PR + CR, of the target lesion, by RECIST 1.1 criteria.
Duration of response | 36 months
  Duration of response by RECIST 1.1
Progression free survival | 36 months
  PFS will be measured from the date of initiation of nab-paclitaxel/paclitaxel plus pembrolizumab to the time of tumor progression or death from any cause
Evaluate the tolerability of radiotherapy added to the combination of chemotherapy and immunotherapy | 36 months
  Adverse events will be assessed according to NCI CTCAE v5.0.
Evaluate change in immune cell populations by IHC. | 36 months
  Serial tumor biopsies will be obtained in a subset of patients and changes in immune cell populations and activation profiles will be evaluated by IHC.
Evaluate change in immune cell populations in blood samples using flow cytometry and gene expression profiling. | 36 months
  Peripheral blood samples will be obtained pre-treatment and at various timepoints after treatment and evaluated by flow cytometry for B cell, NK cell, and CD8, CD4, and regulatory T cell populations including markers of activation and exhaustion (TIM-3, , LAG-3, and PD-L1) and gene expression. Fold change compared to baseline will be determined.
Evaluate changes in markers of immune cell activation using IHC. | 36 months
  Serial tumor biopsies will be obtained in a subset of patients and changes in immune cell populations and activation profiles will be evaluated by IHC.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Diamond, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No